CLINICAL TRIAL: NCT06573944
Title: Intestinal Ultrasound Predicts Upadacitinib Efficacy in Patients With Moderate to Severe Crohn's Disease：a Prospective Study
Brief Title: IUS Predicts Upadacitinib Efficacy in Patients With Moderate to Severe Crohn's Disease：a Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Li Tian, MD, Li Tian,MD[fu3tianli], The Third Xiangya Hospital of Central South University
Other Study IDs: fu3tianli3
Record Dates: First submitted 2024-08-24; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-01

CONDITIONS: Crohn's Disease; Upadacitinib; Intestinal Ultrasound; Predictors
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Crohn's disease (CD) is a chronic nonspecific inflammatory disease of the intestinal tract whose etiology is not yet fully understood, and can present with serious complications such as intestinal obstruction, perforation, abdominal abscesses, and fistulae. Currently, the main therapeutic drugs for CD include aminosalicylic acid preparations, glucocorticoids, immunosuppressants, and biological agents. With the development of medical technology, small molecule preparations have begun to be applied to moderate-to-severe Crohn's disease.

Upadacitinib is a novel oral small molecule agent that is a highly selective JAK-1 inhibitor. A large real-world study showed that in refractory moderate-to-severe CD, upadacitinib showed a clinical response rate of 76.5% and a clinical remission rate of 70.6% at 8 weeks of treatment.

Intestinal ultrasound (IUS) is a noninvasive, reproducible, convenient, and inexpensive test that can greatly increase the frequency of assessing treatment response and speed up the clinical decision-making process.The 2019 ECCO-ESGAR guidelines recommend intestinal ultrasound for disease monitoring in patients with CD. There are no validated indicators to predict the efficacy of upatinib treatment in patients with moderate-to-severe CD in the currently available studies.

Currently, there are no national or international studies in which intestinal ultrasound predicts the efficacy of upatinib therapy. Therefore, we propose for the first time that intestinal ultrasound be used as a method to predict the response to upadacitinib in CD patients, with the aim of providing evidence to guide the development of individualized treatment plans.

DETAILED DESCRIPTION:
Crohn's disease (CD) is a chronic nonspecific inflammatory disease of the intestinal tract whose etiology is not yet fully understood, and can present with serious complications such as intestinal obstruction, perforation, abdominal abscesses, and fistulae. In recent years, the incidence of CD has increased rapidly, causing a heavy social and economic burden. Currently, the main therapeutic drugs for CD include aminosalicylic acid preparations, glucocorticoids, immunosuppressants, and biological agents. With the development of medical technology, small molecule preparations have begun to be applied to moderate-to-severe Crohn's disease, providing new treatment options for patients with moderate-to-severe Crohn's disease. The application of small molecule agents has changed the course of CD. But such drugs need to be taken orally for a long period of time, and there are risks of secondary infections, tumors, and loss of response.So, effective prediction of the efficacy of small molecule agents in patients with moderate-to-severe CD is an urgent clinical problem to be solved.

Upadacitinib is a novel oral small molecule agent that is a highly selective JAK-1 inhibitor. A large real-world study showed that in refractory moderate-to-severe CD, upadacitinib showed a clinical response rate of 76.5% and a clinical remission rate of 70.6% at 8 weeks of treatment. Although upadacitinib offers a new treatment option for patients with refractory moderate-to-severe CD, there are still some patients who have poor outcomes or treatment ineffectiveness with these drugs. Therefore, early screening of patients who respond to upadacitinib and prediction of long-term efficacy are important to guide clinical strategies for CD.

Intestinal ultrasound (IUS) is a noninvasive, reproducible, convenient, and inexpensive test that can greatly increase the frequency of assessing treatment response and speed up the clinical decision-making process.The 2019 ECCO-ESGAR guidelines recommend intestinal ultrasound for disease monitoring in patients with CD. Multiple studies have shown that most ultrasound markers normalize within 12 weeks of treatment initiation, and in particular, normalization of bowel wall thickness is highly correlated with clinical response at 12 weeks. There are no validated indicators to predict the efficacy of upadacitinib treatment in patients with moderate-to-severe CD in the currently available studies.

Currently, there are no national or international studies in which intestinal ultrasound predicts the efficacy of upadacitinib therapy. Therefore, we propose for the first time that intestinal ultrasound be used as a method to predict the response to upadacitinib in CD patients, with the aim of providing evidence to guide the development of individualized treatment plans.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 80 years;
* Patients with newly diagnosed or relapsed moderate to severe Crohn's disease
* Upadacitinib therapy is proposed to be applied within 1 month after baseline endoscopy and intestinal ultrasound,;
* No history of abdominal surgery;
* Clearly understand, voluntarily participate in the study, and sign an informed consent form.

Exclusion Criteria:

* Contraindications to upadacitinib: allergy, active tuberculosis or other active infections, moderate-to-severe heart failure (NYHA grade III/ IV), demyelinating lesions of the nervous system, live vaccination within the last 3 months, pregnancy and lactation;
* Patients with a history of extensive colectomy or recent proposed colectomy, history of colonic mucosal dysplasia;
* Hypersensitivity to the components of SonoVue contrast media.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the Third Xiangya Hospital of Central South University, patients with newly diagnosed or relapsed moderate to severe Crohn's disease treated with upadacitinib will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Bowel wall thickness (BWT) | follow-up time of about 54 weeks
  BWT is measured by intestinal ultrasound. BWT≤3mm means that CD is in quiescent, #3mm means CD is active

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Hunan, Hunan, China

IPD SHARING:
Plan to Share IPD: No
There is not plan to make IPD available